CLINICAL TRIAL: NCT00734890
Title: Phase I Study of Vandetanib (ZD 6474) and Bevacizumab Combination Therapy Evaluating the VEGF and EGF Signal Transduction Pathways in Adults With Solid Tumors and Lymphomas
Brief Title: Vandetanib and Bevacizumab in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 080087; 08-C-0087; NCI-P7189; CDR0000590152
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Lymphoma; Lymphoproliferative Disorder; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; adult nasal type extranodal NK/T-cell lymphoma; Waldenström macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; intraocular lymphoma; post-transplant lymphoproliferative disorder; cutaneous B-cell non-Hodgkin lymphoma; small intestine lymphoma; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; adenosquamous cell lung cancer; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Lung Neoplasms; Lymphoma; Lymphoproliferative Disorders; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Intraocular Lymphoma; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; vandetanib

INTERVENTIONS:
Biological: bevacizumab
Drug: vandetanib
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Vandetanib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bevacizumab and vandetanib may also stop the growth of cancer cells by blocking blood flow to the cancer. Giving vandetanib together with bevacizumab may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vandetanib and bevacizumab in treating patients with advanced solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose, safety, and toxicity of vandetanib and bevacizumab in patients with advanced solid tumors or lymphoma.

Secondary

* Characterize the pharmacokinetic profile of this regimen in these patients.
* Measure changes in VEGF and other angiogenic cytokines in plasma samples from these patients.
* Determine the biochemical changes in the EGF signal transduction pathways in tumor biopsy samples from these patients.
* Determine the anti-angiogenic effects of this regimen in tumor biopsy samples from these patients.
* Evaluate the application of dynamic contrast-enhanced MRI to determine early changes in tumor vascular permeability during treatment.
* Evaluate the effects of this regimen on circulating endothelial progenitors and mature circulating endothelial cells in these patients.

OUTLINE: Patients receive oral vandetanib once daily on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for correlative laboratory studies, including pharmacokinetic, biomarker (VEGF and other angiogenic cytokines), and circulating endothelial cell analysis. Patients may also undergo optional tumor biopsies for additional correlative laboratory studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced malignancy, including the following:

  * Solid tumor that is refractory to standard therapy or for which no standard therapy exists

    * No lung carcinoma of squamous cell or small cell histology (mixed tumors will be categorized by the predominant cell type)

      * Histological confirmation based on sputum cytology alone is not acceptable
  * Lymphoma (Hodgkin or non-Hodgkin lymphoma) that has progressed after standard therapy AND for which stem cell transplantation is not indicated or has been refused
* No known CNS disease, except for treated brain metastasis meeting the following criteria:

  * No ongoing requirement for steroids
  * No evidence of progression or hemorrhage by clinical examination and brain imaging (MRI or CT scan) for ≥ 3 months after treatment

    * Stable dose of anticonvulsants allowed
  * Prior treatment for brain metastases may have included whole-brain radiotherapy, radiosurgery (gamma knife, linear accelerator, or equivalent), or a combination of therapy as deemed appropriate by the treating physician

    * Neurosurgical resection or brain biopsy for treatment of CNS metastases allowed provided treatment was completed more than 3 months ago

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine < 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Urine protein:creatinine ratio ≤ 0.5 OR urine protein < 1,000 mg by 24-hour urine collection
* Activated partial thromboplastin time ≤ 1.5 times ULN
* Prothrombin time OR INR < 1.5 times ULN
* Potassium between 4 mmol/L and ULN (supplementation allowed)
* Magnesium normal (supplementation allowed)
* Serum calcium (adjusted for albumin) or ionized calcium normal (supplementation allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* HIV-positivity allowed provided the following criteria are met:

  * Patient does not require anti-HIV therapy
  * CD4 count > 350/mm^3
  * HIV viral load < 25,000 copies/mm^3
  * No history of opportunistic infections
* No evidence of severe or uncontrolled systemic disease or any concurrent condition that could compromise participation in the study, including any of the following:

  * Active or uncontrolled infection
  * Immune deficiencies
  * HIV infection requiring anti-HIV therapy
  * Hepatitis B
  * Hepatitis C
  * Uncontrolled diabetes
  * Uncontrolled hypertension
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction within the past 6 months
  * Uncontrolled cardiac arrhythmia
  * Stroke/cerebrovascular accident within the past 6 months
  * Psychiatric illness/social situation that, in the investigator's opinion, would make it undesirable for the patient to participate in the study or that would jeopardize study compliance
* No New York Heart Association class III or IV heart disease within the past 6 months
* No history of arrhythmia (i.e., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment

  * Atrial fibrillation allowed provided it is controlled with medication
* No asymptomatic sustained ventricular tachycardia
* No other cardiac disease that, in the investigator's opinion, would increase the risk of ventricular arrhythmia
* QTc < 480 msec (with measurable Bazett correction) by screening ECG
* No history of QTc prolongation as a result of other medications that required discontinuation
* No congenital long QT syndrome
* No first-degree relative with unexplained sudden death at under 40 years of age
* No left bundle branch block
* No hypertension not controlled by medical therapy, defined as systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg despite optimal medical management
* No other clinically significant cardiac event
* No thromboembolic disease within the past 6 months
* No significant vascular disease (e.g., aortic aneurysm or aortic dissection) or clinically significant peripheral vascular disease
* No serious non-healing wounds (including wounds healing by secondary intention)
* No acute or non-healing ulcers
* No bone fractures within the past 3 months
* No abdominal fistula, gastointestinal perforation, or intra-abdominal abscess within the past 28 days
* No currently active diarrhea that may affect the ability of the patient to absorb or tolerate vandetanib
* No hemoptysis (bright red blood of ≥ ½ teaspoon per episode) within the past 3 months
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior anti-VEGF therapy allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy and recovered
* More than 4 weeks since prior major surgery and recovered
* At least 2 weeks since prior investigational drugs given in a phase 0 clinical trial
* More than 10 days since prior and no concurrent aspirin (> 325 mg/day) or chronic use of other NSAIDs
* No concurrent regular, therapeutic anticoagulation
* No concurrent medication that may cause QTc prolongation, induce Torsades de Pointes, or induce CYP3A4 function, including any of the following:

  * Rifampin
  * Rifabutin
  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)
* No other concurrent antineoplastic therapy, except for gonadotropin-releasing hormone therapy for prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Safety
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, MD, Principal Investigator — NCI - Medical Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

REFERENCES:
- [Result] Kummar S, Gutierrez ME, Chen A, Turkbey IB, Allen D, Horneffer YR, Juwara L, Cao L, Yu Y, Kim YS, Trepel J, Chen H, Choyke P, Melillo G, Murgo AJ, Collins J, Doroshow JH. Phase I trial of vandetanib and bevacizumab evaluating the VEGF and EGF signal transduction pathways in adults with solid tumours and lymphomas. Eur J Cancer. 2011 May;47(7):997-1005. doi: 10.1016/j.ejca.2010.12.016. Epub 2011 Jan 17. PMID 21247755